CLINICAL TRIAL: NCT05640583
Title: Assessing the Uniqueness of Inflammatory Bowel Disease Related Microbiome-derived Biomarkers Found in the Lumen of the Human Large Intestine in Comparison to Those Found in Spontaneously Excreted Stool Samples
Brief Title: Assessing Uniqueness of Inflammatory Bowel Disease Related Microbiome-derived Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HyGIeaCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HGP-0011
Record Dates: First submitted 2021-12-18; First posted 2022-12-07 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2021-12

CONDITIONS: Irritable Bowel Disease
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Study Arm = 10 patients diagnosed with colonic IBD (5 diagnosed with Ulcerative Colitis and 5 diagnosed with Crohn's Disease) scheduled for a surveillance colonoscopy
  Control Arm = 10 patients scheduled for a routine screening colonoscopy who do not have a history of IBD symptoms or IBD diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- IBD (Experimental): 10 patients diagnosed with colonic IBD (5 diagnosed with Ulcerative Colitis and 5 diagnosed with Crohn's Disease) scheduled for a surveillance colonoscopy
  Interventions: Device: Hygieacare System
- Control (Active Comparator): 10 patients scheduled for a routine screening colonoscopy who do not have a history of IBD symptoms or IBD diagnosis
  Interventions: Device: Hygieacare System

INTERVENTIONS:
Device: Hygieacare System — The device is an FDA cleared colon irrigation device, it will be used according to clearance. The sampling of the colon effluent sampled is the are of study.

SUMMARY:
To assess the differential expression of IBD-related microbiome-derived biomarkers including bacterial strains and peptides such as antimicrobial peptides (AMP) found in inner-colonic samples (HygiSample™) in comparison to home collected stool samples in patients with active IBD colonic disease.

The HygiSample will be collected during a defecation-inducing high-volume (>40 L) colon irrigation bowel prep (HygiPrepⓇ).

DETAILED DESCRIPTION:
This study is a preliminary study aimed to assess the ability to differentially detect IBD-related microbiome-derived biomarkers in colon effluent samples collected using the Hygieacare System. The proposed sample size of 20 patients (10 in the control arm, 10 in the IBD arm), where each patient provides both stool and three inner-colonic samples is sufficient to provide preliminary results for such an assessment.

Categorical variables will be summarized by frequencies and percentages, while quantitative variables will be summarized by descriptive statistics (mean, median, standard deviation, minimum, and maximum).

The investigators will compare taxonomy and phylogeny biodiversity between the control and the IBD arms and between stool and colon effluent samples.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age is between 18 and 80 years old
* For study arm - patients with known colonic IBD based on colonoscopic findings - diagnosed with either Ulcerative Colitis or Crohn's Disease scheduled for surveillance colonoscopy.
* For control arm - patients scheduled for routine colonoscopy without active IBD symptoms or IBD diagnosis

Exclusion Criteria:

* The patient has an underlying condition that in the opinion of the investigator may adversely affect the patient's ability to understand, comply with, or follow protocol instructions
* History of intestinal resection (appendectomy allowed)
* Active Clostridium difficile colitis
* Antibiotic use for 2 months prior to colonoscopy
* The patient has any of the contraindications listed below:

congestive heart failure, intestinal perforation, carcinoma of the rectum, fissures or fistula, severe hemorrhoids, abdominal hernia, renal insufficiency, cirrhosis, pregnancy, or recent colon, rectal, or abdominal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Detection of IBD-related microbiome-derived biomarkers in stool samples | analysis end of study enrollment
  Each patient provides both stool (when possible) and inner-colonic samples. The samples will be analyzed to identify microorganisms' presence and abundance, diversity, and functional genomics.
  Specifically, we will look at the alpha and beta diversity of the microbiota (% of prediction on the most dominant vectors of the system) and the taxonomic differences between the samples - represented by percentages over taxonomic groups. If the data allows (based on our omics results), we will look at the potential abundance of calprotectin (IBD biomarker, % from control).
  We will analyze the data for the study participants by age, gender, BMI (average, median, standard deviation), and prevalence of underlying diseases.
  The questionnaires will be used to find correlations between the patient's overall health, exercise routine, nutritional habits, and diet. Results will be presented using R^2 when applies.
unpaired T-test | analysis end of study enrollment
  We will track the patients demographic and physiological parameters - age (years), gender (male/female), height (feet inches), weight (lbs), BMI. We will collect information about the patients eating, heath, and exercise habits using a questionnaire.
cox wilcoxon test | through study completion, an average of 1 year
  We will track the patients demographic and physiological parameters - age (years), gender (male/female), height (feet inches), weight (lbs), BMI. We will collect information about the patients eating, heath, and exercise habits using a questionnaire

SECONDARY OUTCOMES:
Differential abundance analysis | through study completion, an average of 1 year
  For our comparative analyses, we will carry out clustering and differential abundance. we will qualify the bacteria abundance using 16S and meta genomics analysis and provide information of the available species using Alpha diversity and Shannon index and beta diversity using PCoA analysis.
  analysis with correction for multiple comparisons by false discovery rate.
Alpha diversity | through study completion, an average of 1 year
  16S and meta genomics analysis
Shannon index | through study completion, an average of 1 year
  16S and meta genomics analysis
beta diversity | through study completion, an average of 1 year
  PCoA analysis

CONTACTS AND LOCATIONS:
Overall Officials: David A Johnson, MD, Principal Investigator — Digestive & Liver Disease Specialists
Locations (1):
- Hygieacare Center, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The outcome of the colon effluent analysis will be published.